CLINICAL TRIAL: NCT07147673
Title: Brain Function During Grasping Task in Three to Nine Months Infants Using fNIRS , the Difference Between Full and Preterm Born Infants
Brief Title: fNIRS Grasping Task in Infants
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0265
Record Dates: First submitted 2025-04-14; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Preterm and Term Infants
Keywords: fNIRS; grasping; infants; preterm infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- full term infants: infants between 3-9 months old with gestational age more than 36 weeks
- preterm infants: infants between 3-9 months old corrected age born with a gestational age less than 36 weeks

SUMMARY:
This study aims to investigate the neural mechanisms involved in the development of reach-to-grasp function in infants. Reaching and grasping are crucial motor skills that develop early in infancy and are essential for later motor and cognitive milestones. Understanding how these skills emerge and the underlying neural processes can provide valuable insights into both typical and atypical development.

The study will focus on infants aged 3 to 9 months, a critical period for the development of reach-to-grasp skills. A total of 100 infants will be recruited, including 50 full-term infants and 50 preterm infants (born <36 weeks gestational age). Reach-to-grasp function will be evaluated through a cross-sectional assessment at a single time point. Functional near-infrared spectroscopy (fNIRS) will be used as the brain imaging technique to measure brain activity during the reach-to-grasp task. The use of fNIRS will allow for a non-invasive assessment of neural activity in real time, providing insights into the brain mechanisms supporting the development of motor skills. The findings may offer important information about the neural basis of motor development in infancy, particularly in the context of preterm birth.

DETAILED DESCRIPTION:
This study aims to investigate the neural mechanisms underlying the development of grasping function in infants aged 3 to 9 months. Specifically, it focuses on brain activity linked to reach-to-grasp movements, the role of maturation in this brain activity, the effect of preterm birth, and brain activity during bimanual toy exploration. The study will recruit 100 infants, including 50 full-term infants and 50 preterm infants (born at less than 36 weeks gestational age). Functional Near-Infrared Spectroscopy (fNIRS) will be used as the brain imaging technique to assess neural activity.

Objectives:

To investigate differences in brain activity during the reach-to-grasp task in 3-9-month-old infants between preterm and full-term infants.

To evaluate differences in the neural correlates of maturation of the reach-to-grasp motor skill.

To investigate differences in laterality index between preterm and full-term infants during bimanual toy exploration.

Method:

Fifty preterm and fifty full-term infants between 3 and 9 months corrected age will be assessed at a single time point. The assessment consists of an fNIRS event-related reach-to-grasp task protocol, where infants are encouraged to reach and grasp a toy, measured using the NSP2 system (NIRx). The task protocol includes 10 repetitions of each reach-to-grasp condition: 5 seconds of left-hand reach-to-grasp, 5 seconds of right-hand reach-to-grasp, and 10 seconds of bimanual toy exploration. A 10-second rest period is implemented between each reach-to-grasp action, and a 30-second rest period is implemented between conditions. Additionally, 5-7 minutes of resting-state fNIRS data will be recorded while infants watch a screensaver-like video to help maintain a resting state.

The fNIRS cap configuration consists of an 8×8 optode array covering the sensorimotor cortex. Cap size is adapted to the infant's head circumference (ranging between 42 and 46 cm), with the optode configuration remaining consistent across all cap sizes.

In addition to the fNIRS assessment, two clinical assessments will be conducted:

Hand Assessment for Infants (HAI): Evaluates hand function in infants. Hammersmith Infant Neurological Examination (HINE): Assesses neurological development.

ELIGIBILITY:
Inclusion Criteria:

* 3-9 months old
* can tolerate the fNIRS cap
* performs at least 2 grapsing attempts with one hand within one minute when prompting the hand with a toy

Exclusion Criteria:

* history of periferal neurological lesion such as plexus brachialis lesion
* presence of epilepsia, congenital brain malformation,
* no informed consent
* severe visual impairments
* syndromal or genetical diseases resulting into developmental delay

Ages: 3 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infants between 3 an 9 months old, living in Flanders (Belgium) born full term or preterm.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
fNIRS laterality index | Baseline
  Difference in brain activitity over the sensorimotor cortex between left and right hemisphere during bilateral grasping. Averaged brain activity of the 10 blocks of bimanual grasping.

SECONDARY OUTCOMES:
fNIRS bimanual activity | baseline
  Averaged brain activity during the 10 blocks of bimanual reach-to-grasp movements.
fNIRS unmanual left-sided activity | baseline
  Averaged brain activity during the 10 blocks of unilateral left-sided reach-to-grasp movements.
Hand assessment for Infants (HAI) | baseline
  An assessment of hand function. It has been developed for infants at risk of developing cerebral palsy (CP) in the age range of 3-12 months. The HAI intends to measure the degree and quality of goal directed actions performed with each hand separately as well as with both hands together.
  Items are scored based on a video-taped play session eliciting upper limb activity.
  It results in three scales
  1. both hand measure: a criterian referenced overall measure of hand function based on all 17 items total raw score ranges ; 0-58 HAI-unit scale: 0-100 Higher score indicates better ability
  2. each hand sum score: a unimanual criterion referenced subscale based on 12 out of 17 items, score rated for each hand seperatly raw score ranges: 0-24 higher score indicates better ability
  3. percentage of difference between hands : percent calculated by the differences in left and right each hand sum score higer value indicate bigger difference between hands
  age norm references available
Hammersmith infant neurological examination (HINE) | baseline
  Hammersmith infant neurological examniation is a standardized neurological exam for infants adjusted age 2 to 24 months. The HINE evaluates nerve function, movements, reflexes and reactions, posture, and tone and can help clinicians identify movement disorders including cerebral palsy (CP).
  26 items scoring 0-3 total score : 0-78 Higher score indicates more optimal developement normative data for age-matched, typically developing infants helps determine if the score is optimal or suboptimal.
fNIRS resting state functional connectivity | baseline
  Functional connectivity within the sensorimotor cortex during a 5-7minutes of rest.
fNIRS unmanual right-sided activity | baseline
  Averaged brain activity during the 10 blocks of unilateral right-sided reach-to-grasp movements.

CONTACTS AND LOCATIONS:
Overall Officials: Nele De Bruyn, Phd, Principal Investigator — University Ghent
Locations (1):
- hent University, vakgroep revalidatiewetenschappen, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
It concerns personal data. There must first be investigated to which extent this data can be pseunominized for sharing.